CLINICAL TRIAL: NCT02164903
Title: Mid to Long-term Quality of Life Effects Of imatiNIb Versus DASatinib in Chronic Myeloid Leukemia Patients (LEONIDAS)
Brief Title: LEONIDAS: Quality of Life Study in Chronic Myeloid Leukemia Patients
Acronym: QoL-CML0713
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Collaborators: European Leukemia Net (Unknown); CML Advocates Network (Unknown)
Responsible Party: Sponsor
Other Study IDs: QoL-CML0713
Record Dates: First submitted 2014-05-27; First posted 2014-06-17 (Estimated); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Chronic Myeloid Leukemia
Keywords: Quality of Life; Chronic Myeloid Leukemia; Imatinib; Dasatinib
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Imatinib: Patients in first line treatment with imatinib for no more than 3 years.
  Interventions: Other: QoL Survey Booklet
- Dasatinib: Patients in first line treatment with dasatinib for no more than 3 years.
  Interventions: Other: QoL Survey Booklet

INTERVENTIONS:
Other: QoL Survey Booklet

SUMMARY:
The broad goal of this study is to investigate if differences exist (and in which areas and of what magnitude) in QoL and symptoms of patients with CML being treated with first line therapy with dasatinib versus those receiving first line therapy with imatinib. Also, an additional objective is to characterize medication-taking behavior associated with imatinib or dasatinib.

DETAILED DESCRIPTION:
The development of molecular targeted therapies (i.e., oral tyrosine kinase inhibitors [TKIs]) to treat chronic myeloid leukemia (CML) is one of the great triumphs of modern oncology and one of the spearheads of personalized medicine. Since their introduction in 2001, the number of people living with CML has doubled, a trend that is expected to continue.

This study (i.e., LEONIDAS) is set up to generate evidence-based data and produce information that will advance scientific knowledge, clinical practice and health services management to facilitate clinical decision-making in CML.

In an effort to further promote patient-centered care for CML a patient advocacy organization, that is the: CML Advocates Network, is involved in this project with key representatives who will be in the advisory board team. The CML Advocates Network, hosted by the patient-run, non-profit Leukemia Patient Advocates Foundation is a worldwide network of 82 non-profit organizations from 63 countries supporting patients with CML and their relatives.

Rationale and Significance Some ten years ago, the treatment of CML was relatively straightforward as all patients received imatinib as first-line treatment and for those who failed imatinib, the only available proven alternative was allogeneic stem cell transplantation. Nowadays, with three effective drugs (i.e., imatinib, nilotinib and dasatinib), that can be used frontline in newly diagnosed chronic phase (CP) CML patients, treatment decision-making for individual patients in daily clinical practice has thus rapidly grown in complexity. Moreover, a new tyrosine kinase inhibitors (TKI), bosutinib, has been recently approved for as second-line treatment and undergoing clinical trials are assessing its efficacy as frontline strategy in CML.

To further complicate the scenario, is the fact that despite nilotinib and dasatinib have been shown to have higher rates of cytogenetic and molecular responses (compared to imatinib), none of these three drugs is dramatically better than the others. To illustrate, only slightly differences exist in terms of progression-free survival for nilotinib and no differences for overall survival at 24 and/or 36 months amongst imatinib, dasatinib and nilotinib.

Nevertheless, physician-reported toxicity data suggests these drugs have different toxicity profiles, with imatinib inducing a higher proportion of low-grade side effects than second generation tyrosine kinase inhibitors (TKI) (i.e. nilotinib and dasatinib).

While a wealth of biomedical and laboratory data exists on clinical efficacy of these three drugs, the impact of these from the patients' perspective, in terms of Quality of Life (QoL) and symptom burden, has been poorly investigated. No data exists on QoL of patients treated with nilotinib or dasatinib and it is not known if these drugs provide better QoL outcomes over imatinib when used as first line therapy. Such information would be critical in the current CML arena to make more informed treatment decisions. This is a significant gap in our knowledge with respect to the modern management of CML, also because, as long-term continuous exposure to the tyrosine kinase inhibitors (TKI) is necessary, even low grade side effects can heavily impact on patients' QoL.

Thus, the objective of this study is to investigate if differences exist (and in which areas and of what magnitude) in QoL and symptoms of patients with CML being treated with first line therapy with dasatinib versus those receiving first line therapy with imatinib, as well as characterizing medication-taking behavior associated with imatinib or dasatinib.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older at the time of study entry;
* Diagnosis of Philadelphia chromosome positive and/or BCR-ABL positive CML confirmed by cytogenetic and/or molecular analysis;
* At least in CCyR (as documented by chromosome banding analysis of marrow cell metaphases) or in MMR (≤0.1% BCR-ABL IS)
* CP-CML Patients in first line treatment with either dasatinib or imatinib for no more than 3 years;
* Written informed consent.

Exclusion Criteria:

* Major cognitive deficits or psychiatric problems hampering a self-reported evaluation.
* Not speaking and reading the language of the participating country.
* Having received any CML treatment prior to therapy with imatinib or dasatinib for more than three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult chronic myeloid leukemia patients in first line treatment with either dasatinib or imatinib for no more than 3 years.
Sampling Method: Non-Probability Sample
Enrollment: 323 (Actual)
Dates: Start 2014-09-11 (Actual); Primary Completion 2017-01-25 (Actual); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Severity of the impact of therapy on daily life in patients with CP-CML being treated with first line therapy with dasatinib and those receiving first line therapy with imatinib. | 24 months.
  (outcome measure: European Organization for Research and EORTC QLQ-CML24 "Impact on daily life" scale)

SECONDARY OUTCOMES:
Differences in Patient-reported outcomes between imatinib- and dasatinib- treated CP- CML patients in the following QoL domains: Fatigue, Physical, Social and Role Functioning and Impact on worry and mood and Symptom burden. | 24 months.
  (outcome measure: EORTC QLQ-C30 and EORTC QLQ-CML24)
Proportion of patients considered as low, medium and high adheres by type of therapy. | 24 months.
  (outcome measure: Morisky-Medication Adherence Scale-MMAS)
Relationship between patient's perception of disease-/treatment-related information received , QoL profile and adherence to therapy. | 24 months.
  (defined according to the EORTC-QLQ-INFO25)
Degree of agreement in the assessment of symptom severity, for a set of core CML treatment related symptoms , between patients and their treating physicians. | 24 months.
  (according to the EORTC-QLQ-CML24)

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Efficace, PhD, Study Chair — Gruppo Italiano Malattie EMatologiche dell'Adulto; Gianantonio Rosti, Dr., Study Director — University of Bologna
Locations (49):
- Department of Hematology and Oncology, Hôpital Mignot, Université Versailles Saint-Quentin-en-Yvelines, Le Chesnay, France
- Germany (2):
  - Universität Heidelberg - III. Medizinische Klinik - Universitätsmedizin Mannheim, Mannheim
  - Universitat Heidelberg, Mannhein
- Italy (45):
  - S. C. di Ematologia - Azienda Ospedaliera - SS. Antonio e Biagio e Cesare Arrigo, Alessandria
  - Clinica di Ematologia - Azienda Ospedaliera Regionale di Torrette, Ancona
  - U.O. Ematologia con trapianto - Azienda Ospedaliero-Universitaria Policlinico di Bari, Bari
  - Istituto di Ematologia "L. e A. Seragnoli" - Università degli Studi di Bologna - Policlinico S. Orsola - Malpighi, Bologna
  - USD - Centro Trapianti Midollo Osseo Adulti - Cattedra di Ematologia - Azienda Spedali Civili - Brescia, Brescia
  - U.O. Ematologia Brindisi- Ospedale A. Perrino ASL BR, Brindisi
  - CTMO-Ematologia-Ospedale "Binaghi", Cagliari
  - U.O. Ematologia CTMO "Businco", Cagliary
  - Divisione clinicizzata di Ematologia - Dipartimento di Scienze Mediche - Osp. Ferrarotto, Catania
  - Azienda Ospedaliera - Arcispedale S. Anna Sezione di Ematologia e Fisiopatologia delle Emostasi, Ferrara
  - Divisione di Ematologia - Policlinico Careggi, Florence
  - Clinica Ematologica - Dipartimento di Medicina Interna - IRCCS San Martino - IST, Genova
  - Divisione di Ematologia - Azienda Ospedaliera Ospedali Riuniti "Papardo Piemonte", Messina
  - Divisione Ematologia - Dipartimento di Medicina Interna -Policlinico Universitario di Messina, Messina
  - U.O. Ematologia - Azienda USLL12 Veneziana - Ospedale dell'Angelo e Ospedale civile S. Giovanni e Paolo, Mestre - Venezia
  - U.O. Ematologia 1 - Centro Trapianti di Midollo - Ospedale Maggiore Milano, Milan
  - Dipartimento di Med. Clinica e Sperimentale- Area di Ematologia - Facoltà di Medicina e Chirurgia - Università degli Studi di Napoli "Federico II" -, Napoli
  - U.O. Ematologia - Ospedale S. Gennaro, Napoli
  - XIX Divisione di Ematologia con trapianto - A.O.R.N. "A. Cardarelli", Napoli
  - Divisione di Ematologia - Dip. Di Medicina Clinica e Sperimentale & BRMA - Università Piemonte Orientale "Amedeo Avogato", Novara
  - Dipartimento di Scienze Cliniche e Biologiche - Ospedale S. Luigi Gonzaga, Orbassano
  - Ematologia ed Immunologia Clinica - Università degli studi di Padova, Padua
  - Divisione di Ematologia con trapianto di midollo - A.O.U. Policlinico "Paolo Giaccone", Palermo
  - U.O.C. Ematologia - A.O. Ospedali Riuniti "Villa Sofia-Cervello", Palermo
  - Ematologia e CTMO - A.O.U. Università degli Studi di Parma, Parma
  - Unità Operativa Ematologia e Centro Trapianti - Dipartimento di Oncologia ed Ematologia - AUSL Ospedale di Piacenza, Piacenza
  - U.O. Ematologia - A.O.U. Pisana, Pisa
  - U.O. Ematologia - A.O. San Carlo, Potenza
  - Divisione di Ematologia - A.O. Ospedali Riuniti di Reggio Calabria "Bianchi-Melacrino-Morelli", Reggio Calabria
  - Rimini Ospedale "Infermi", Rimini
  - Department of Onco-Hematology - IRCCS; Centro di Riferimento Oncologico della Basilicata, Rionero in Vulture
  - Clinica di Ematologia - Policlinico Umberto I- Università degli Studi "Sapienza", Roma
  - Divisione di Ematologia - Ospedale S.Eugenio, Roma
  - Ematologia - A.O. Sant'Andrea, Roma
  - Ematologia Policlinico - Università degli Studi di Roma Tor Vergata (PTV), Roma
  - U.O. di Ematologia - Ente Ospedaliero San Giovanni Addolorata, Roma
  - U.O.C. Ematologia e Trapianto cellule staminali - Pad Cesalpino- A.O. San Camillo Forlanini, Roma
  - U.O. di Ematologia - Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - Ematologia - AOU Sassari, Sassari
  - U.O.C. Ematologia - A.O. SS Annunziata - P.O.S.G. Moscati, Taranto
  - S.C. di Oncoematologia - A.O. "S. Maria", Terni
  - S.C.D.O. Ematologia II - A.O.U.S. San Giovanni Battista di Torino (Molinette), Torino
  - Clinica Ematologica ed Unità di Terapie Cellulari Carlo Melzi - A.O. Universitaria, Udine
  - Onco-Ematologia - Ospedale S. Andrea- Vercelli, Vercelli
  - U.O di Ematologia d. U. - Azienda Ospedaliera Universitaria Integrata Verona, Verona
- Department of Hematology, Hospital Universitario de la Princesa, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gruppo Italiano Malattie EMatologiche dell'Adulto (GIMEMA) Foundation — http://www.gimema.it